CLINICAL TRIAL: NCT02202278
Title: Serum Levels of IMA, TAC, TOS, OSI and MDA in Severe OHSS Patients Underwent Long Agonist Protocol Intracytoplasmic Sperm for Determining Oxidative Stress Status
Brief Title: Study of Serum Levels of Oxidative Stress Markers in Ovarian Hyperstimulation Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, emine seda guvendag guven, medical doctor, Karadeniz Technical University
Other Study IDs: 139EK1
Record Dates: First submitted 2014-07-23; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: ovarian hyperstimulation; Oxidative Stress; IMA; OHSS; ICSI; long agonist protocol; TAC; TOS; OSI; MDA
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood of involved patients in study was drawn for study for ischemia modified albumin (IMA), malondialdehyde (MDA), total oxidative capacity (TOS), total antioxidative capacity (TAS) and oxidative stress capacity (OSI) levels. After the study all blood samples will be destroyed according to regulations.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ovarian hyperstimulation patients: Moderate OHSS is defined as abdominal distension and discomfort, nausea with or without vomiting, ovarian enlargement (ovarian size of 8-12 cm) and ascites that revealed by ultrasonografic examination. Severe OHSS criteria is defined as ovarian enlargement, ascites with or without hydrothorax, haematocrit >45%, weight gain >2 kg, white blood cell count >15.000, oliguria, creatinine of 1.0-1.5, creatinine clearance of >50 ml/min, liver dysfunction.
- without ovarian hiperstimulation: Control group is composed of patients who underwent long luteal protocol but do not demonstrate symptoms of OHSS

SUMMARY:
The aim of the study is to determine serum oxidative stress status by ischemia modified albumin (IMA), total antioxidant capacity (TAC), total oxidative capacity (TOS), oxidative stress capacity (OSI), and serum malondialdehyde (MDA) in patients with OHHS and control group. We also aim to reveal the association between serum levels of these factors and oocyte quality.

DETAILED DESCRIPTION:
* Patients included in this study were assisted reproductive technique (ART) patients with moderate and severe OHSS who were hospitalized for management
* Control patients are selected from patients without signs of OHSS
* All patients are administered luteal long protocol for controlled ovarian stimulation. Pituitary down-regulation with SC injection of GnRH agonist (GnRH-a) (1 mg/day; Lucrin, Abbott Laboratories, North Chicago, IL) that was started on day 21 of the previous menstrual cycle. Subcutaneous administration of recombinant hFSH (Gonal-F, Laboratories Serono S.A., Aubonne, Switzerland) at dosages from 150-225 IU/day is initiated on the second or third day of menstruation.
* When there are at least two or three follicles >17 mm in diameter, recombinant human chorionic gonadotropin (0.25 µgr ; Ovitrelle IM, Serono, Istanbul, Turkey) is applied subcutaneously 34-36 hours before oocyte retrieval.
* Serum samples are collected on day of HCG for study and control group patients.
* Serum levels of ischemia modified albumin (IMA), malondialdehyde (MDA), total oxidative capacity (TOS), total antioxidative capacity (TAS) and oxidative stress capacity (OSI) levels.
* This is a case control study
* Statistical analyses will be performed using student t-test and fisher chi-square test. The correlations between the serums IMA, TAC, TOC, OSI, and MDA levels will be examined in all study groups using Spearman correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

• Patients in both groups are normoresponders or hyperresponders who will undergo assisted reproductive technology for male factor

Exclusion Criteria:

* known inherited or acquired thrombophilia
* previous thromboembolism
* previous, current or planned anti-thrombotic treatment
* first degree relatives with known genetic thrombophilia
* systemic diseases
* smoking.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients that are administered luteal long protocol for controlled ovarian stimulation
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change the levels of oxidative stress markers | 1 day
  Serum will be obtained for studiying ischemia modified albumin (IMA), malondialdehyde (MDA), total oxidative capacity (TOS), total antioxidative capacity (TAS) and oxidative stress capacity (OSI) levels

CONTACTS AND LOCATIONS:
Overall Officials: emine seda guvendag guven, MD, Study Director — Karadeniz Technical University; rafet duraker, MD, Principal Investigator — T. C Etlik Zubeyde Hanim Women's health Teaching Hospital
Locations (1):
- T.C Saglik Bakanligi Etlik Zübeyde Hanim Womens Health Teaching Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Hitkari JA, Rowe TP, von Dadelszen P. Activated protein C and the ovarian hyperstimulation syndrome: possible therapeutic implications. Med Hypotheses. 2006;66(5):929-33. doi: 10.1016/j.mehy.2005.08.058. Epub 2006 Jan 24. PMID 16434147
- [Background] Westerlund E, Henriksson P, Wallen H, Hovatta O, Wallberg KR, Antovic A. Detection of a procoagulable state during controlled ovarian hyperstimulation for in vitro fertilization with global assays of haemostasis. Thromb Res. 2012 Oct;130(4):649-53. doi: 10.1016/j.thromres.2011.11.024. Epub 2011 Dec 7. PMID 22154245
- [Background] Agarwal A, Allamaneni SS. Role of free radicals in female reproductive diseases and assisted reproduction. Reprod Biomed Online. 2004 Sep;9(3):338-47. doi: 10.1016/s1472-6483(10)62151-7. PMID 15353087
- [Background] Velthut A, Zilmer M, Zilmer K, Kaart T, Karro H, Salumets A. Elevated blood plasma antioxidant status is favourable for achieving IVF/ICSI pregnancy. Reprod Biomed Online. 2013 Apr;26(4):345-52. doi: 10.1016/j.rbmo.2012.12.012. Epub 2013 Jan 16. PMID 23415995